CLINICAL TRIAL: NCT06970847
Title: 64Cu-SAR-bisPSMA Positron Emission Tomography: A Phase 3 Study of Participants With Biochemical Recurrence of Prostate Cancer
Acronym: AMPLIFY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Clarity Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLP10
Record Dates: First submitted 2025-04-29; First posted 2025-05-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Prostate Cancer Patients With Detectable PSA Following Prostatectomy; Prostate Cancer Recurrent; Prostate Cancer Patients Who Have Brachytherapy Seed Implant; Prostate Cancer Patients Treated by Radiotherapy; Cryotherapy
Keywords: Prostate Cancer; Prostate; Biochemical Recurrence
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 64Cu-SAR-bisPSMA 200MBq 64Cu-SAR-bisPSMA. (Experimental)
  Interventions: Drug: 64Cu-SAR-bisPSMA

INTERVENTIONS:
Drug: 64Cu-SAR-bisPSMA — All Patients will receive a single administration, a bolus injection of 200MBq 64Cu-SAR-bisPSMA

SUMMARY:
The aim for this study is to investigate the ability of 64Cu-SAR-bisPSMA PET/CT to detect recurrence of prostate cancer

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Signed informed consent.
3. Life expectancy ≥ 6 months as determined by the Investigator.
4. Histologically confirmed adenocarcinoma of prostate per original diagnosis and completed subsequent definitive therapy.
5. Participant potentially eligible for salvage therapy with curative intent (i.e. aligns with the definition of loco-regional therapy as described in protocol Section 7.2).
6. PSA level after definitive therapy:

   1. Post-radical prostatectomy: Detectable or rising PSA that is ≥ 0.2 ng/mL with a confirmatory PSA ≥ 0.2 ng/mL (per AUA recommendation) or
   2. Post-radiation therapy, cryotherapy, or brachytherapy: Increase in PSA level that is elevated by ≥ 2 ng/mL above the nadir (per ASTRO-Phoenix consensus definition).
7. Participant willing to undergo biopsy of a 64Cu-SAR-bisPSMA PET-positive lesion for histological confirmation of PC, where this is safe and feasible.
8. An Eastern Cooperative Oncology performance status of 0-2.

Exclusion Criteria:

1. Participants who received investigational agent within 5 biological half-lives prior to Day 1.
2. Participants administered any high energy (>300 KeV) gamma-emitting radioisotope within 5 physical half-lives prior to Day 1.
3. Participants with known predominant small cell or neuroendocrine PC.
4. Previous systemic therapy for PC (with the exception of neoadjuvant and adjuvant systemic therapy as part of the definitive therapy and/or salvage therapy with radiation).
5. Ongoing treatment or treatment within 6 months of Day 1 with any systemic therapy (e.g. any investigational therapy, androgen-deprivation therapy, antiandrogen, gonadotropin-releasing hormone, luteinizing hormone-releasing hormone agonist or antagonist, chemotherapy, immunotherapy or radiotherapy) for PC.
6. Participants for whom there is an intent to initiate a prohibited medication(s)/treatment(s) (refer to Section 7.3) during the course of the participant's involvement in the study.
7. Known or expected hypersensitivity to 64Cu-SAR-bisPSMA or any of its components.
8. Any serious medical condition or extenuating circumstance (including receiving the investigational product or not capable of having a PET scan) which the investigator feels may interfere with the procedures or evaluations of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Ability of 64Cu-SAR-bisPSMA PET/CT to detect recurrence of prostate cancer | Up to 52 Weeks
  Co-primary endpoints of participant-level CDR and region level PPV assessed independently for Day 1 and Day 2:
  * Participant-level CDR, defined as the proportion of TP participants scan out of all participants
  * Region-level PPV, defined as the proportion of TP regions out of all positive regions.

SECONDARY OUTCOMES:
To investigate the safety and tolerability of 64-CuSAR-bisPSMA | Up to 52 Weeks
  Incidence and severity of TEAEs and SAEs following the administration of 64CuSARbisPSMA
To assess the participants-level PPV of 64Cu-SAR-bisPSMA PET/CT | Up to 52 Weeks
  Participant-level PPV, defined as the proportion of participants with a TP scan out of all participants with a true or false positive scan.
To assess the participant-level DR of 64Cu-SAR-bisPSMA PET/CT | Up to 52 Weeks
  Participant-level DR, defined as the proportion of participants with a positive scan out of all participants.
To determine the efficacy of 64Cu-SAR-bisPSMA PET/CT in participants with negative or equivocal conventional imaging at baseline | Up to 52 Weeks
  Detection Rate in participants with a negative or equivocal conventional imaging at baseline.
To determine the effect of the composition of Reference Standard on the performance of 64Cu-SAR-bisPSMA PET/CT | Up to 52 Weeks
  Positive Predictive Value (participant- and region-level) assessed in subgroups based on the type of evidence and with/without histopathology.
To evaluate the consistency among readers and the reproducibility of the 64Cu-SAR-bisPSMA PET/CT readings | Up to 52 Weeks
  Inter-reader variability expressed with kappa statistics for the 64Cu-SAR-bisPSMA PET/CT interpretation by the three central readers.
To evaluate the consistency among readers and the reproducibility of the 64Cu-SAR-bisPSMA PET/CT readings | Up to 52 Weeks
  Intra-reader variability expressed with kappa statistics for the 64Cu-SAR-bisPSMA PET/CT interpretation by the three central readers.
To determine the efficacy of 64Cu-SAR-bisPSMA PET/CT in participants with negative or equivocal conventional imaging at baseline | Up to 52 Weeks
  Positive Predictive Values (participant and region level) in participants with a negative or equivocal conventional imaging at baseline.
To determine the effect of the composition of Reference Standard on the performance of 64Cu-SAR-bisPSMA PET/CT | Up to 52 Weeks
  Correct Detection Rate assessed in subgroups based on the type of evidence and with/without histopathology.

CONTACTS AND LOCATIONS:
Locations (27):
- United States (23):
  - East Valley Urology Center of Arizona, Mesa, Arizona
  - Arkansas Urology Research Center, Little Rock, Arkansas
  - UC Irvine, Irvine, California
  - Comprehensive Urology Medical Group, Los Angeles, California
  - Alarcon Urology Center, Montebello, California
  - University of Florida Health- Jacksonville, Jacksonville, Florida
  - Biogenix Molecular, Miami, Florida
  - Endeavor Health, Evanston, Illinois
  - Indiana University Health-IU Simon Cancer Center, Indianapolis, Indiana
  - Wichita Urology Group, Wichita, Kansas
  - XCancer Research Network / LCMC Health EJGH, Metairie, Louisiana
  - St. Louis University, St Louis, Missouri
  - XCancer, Omaha, Nebraska
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
  - Houston Metro Urology-SW, Houston, Texas
  - The Urology Place, San Antonio, Texas
  - Summit Urology, Murray, Utah
  - Intermountain Medical Center, Salt Lake City, Utah
- Australia (4):
  - St. Vincent's Hospital, Sydney, Darlinghurst, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Westmead Private Hosptial, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland

IPD SHARING:
Plan to Share IPD: No
Concerns related to confidentiality.